CLINICAL TRIAL: NCT05368025
Title: Staying Connected: a Mobile Health Study for Remote Monitoring of Dysphagia Exercises and Patient-reported Outcome Measures
Brief Title: Staying Connected: a Mobile Health Study With the Noona® and Mobili-T® Systems
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00094960
Record Dates: First submitted 2022-02-15; First posted 2022-05-10 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Newly diagnosed Oropharyngeal cancer patients: Newly diagnosed oropharyngeal cancer patients will be enrolled into the study. Patients will receive both mobile health systems and be asked to complete swallowing exercises and report symptoms daily for a period of 6 months. Following completion of the study, this group will be interviewed individually to gain insight into the user experience of using both systems
  Interventions: Device: Mobili-T/Noona

INTERVENTIONS:
Device: Mobili-T/Noona — Use of two mobile health systems over a period of 6 months

SUMMARY:
Mobile health applications are an attractive technological solution that facilitates access to care for patients conveniently and efficiently. Research has shown that remote mHealth delivery has improved patient reported outcomes of disease severity. While such outcomes have traditionally been collected at one point in time within a clinical setting, the potential exists to now gather patient perspectives remotely. Additionally, when combined with a mobile health device, mHealth apps can objectively monitor a treatment plan.

Before implementing a new technology, it is important to investigate how digital health technologies are best integrated into clinical workflows, and how more than one technology can work together to streamline the process. Additionally, it is important to understand the relative benefits of each system from a user perspective and identify how combined data can benefit clinical workflows. Therefore, the purposes of this project are to demonstrate how two technology companies can work together to assess the feasibility of implementing two related systems into one care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of head and neck cancer;
* Will be receiving treatment for head and neck cancer (e.g., +/-surgery, +/- radiation therapy, +/- chemotherapy);
* The primary site of their cancer is the oropharynx, as this is the subgroup of patients known to experience dysphagia.

Exclusion Criteria:

* Have a history of cognitive delay,
* History of stroke or traumatic brain injury.
* Have a beard that they are not willing to shave or partially shave (as the device adheres under the chin, on the surface of the skin).
* Have an implanted electronic device of any kind, including cardiac pacemakers or similar assistive devices, electronic infusion pumps, and implanted stimulators
* Have irritated skin or skin with open wounds under the chin;
* Have an allergy to silver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed Oropharyngeal Cancer patients
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
The MD Anderson Dysphagia Inventory (MDADI) to assess dysphagia severity in those with a history of HNC | pre-operative
  The MD Anderson Dysphagia Inventory (MDADI) is a validated and reliable self-administered questionnaire that was specifically designed for patients with a history of HNC. MDADI consists of 20 questions and results in 4 subscales: global, emotional, functional and physical. Although no gold standard questionnaire exists for HNC patients, a recent systematic review revealed that MDADI was one of the most frequently utilized and thoroughly tested instruments for symptom-specific HNC measures. While all subscores will be reported for demographic purposes, only the composite score will be used for statistical analyses.
The MD Anderson Dysphagia Inventory (MDADI) to assess dysphagia severity in those with a history of HNC | 1 month post-surgery
  The MD Anderson Dysphagia Inventory (MDADI) is a validated and reliable self-administered questionnaire that was specifically designed for patients with a history of HNC. MDADI consists of 20 questions and results in 4 subscales: global, emotional, functional and physical. Although no gold standard questionnaire exists for HNC patients, a recent systematic review revealed that MDADI was one of the most frequently utilized and thoroughly tested instruments for symptom-specific HNC measures. While all subscores will be reported for demographic purposes, only the composite score will be used for statistical analyses.
The MD Anderson Dysphagia Inventory (MDADI) to assess dysphagia severity in those with a history of HNC | 3 months post-surgery
  The MD Anderson Dysphagia Inventory (MDADI) is a validated and reliable self-administered questionnaire that was specifically designed for patients with a history of HNC. MDADI consists of 20 questions and results in 4 subscales: global, emotional, functional and physical. Although no gold standard questionnaire exists for HNC patients, a recent systematic review revealed that MDADI was one of the most frequently utilized and thoroughly tested instruments for symptom-specific HNC measures. While all subscores will be reported for demographic purposes, only the composite score will be used for statistical analyses.
The MD Anderson Dysphagia Inventory (MDADI) to assess dysphagia severity in those with a history of HNC | 6 months post-surgery
  The MD Anderson Dysphagia Inventory (MDADI) is a validated and reliable self-administered questionnaire that was specifically designed for patients with a history of HNC. MDADI consists of 20 questions and results in 4 subscales: global, emotional, functional and physical. Although no gold standard questionnaire exists for HNC patients, a recent systematic review revealed that MDADI was one of the most frequently utilized and thoroughly tested instruments for symptom-specific HNC measures. While all subscores will be reported for demographic purposes, only the composite score will be used for statistical analyses.
The Health Questionnaire (EuroQoL EQ-5D) will assess health status in terms of five dimensions of health | pre-operative
  The Health Questionnaire (EuroQoL EQ-5D) will be administered. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. The 5 areas that it measures include: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
The Health Questionnaire (EuroQoL EQ-5D) will assess health status in terms of five dimensions of health | 1 month post-surgery
  The Health Questionnaire (EuroQoL EQ-5D) will be administered. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. The 5 areas that it measures include: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
The Health Questionnaire (EuroQoL EQ-5D) will assess health status in terms of five dimensions of health | 3 months post-surgery
  The Health Questionnaire (EuroQoL EQ-5D) will be administered. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. The 5 areas that it measures include: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
The Health Questionnaire (EuroQoL EQ-5D) will assess health status in terms of five dimensions of health | 6 months post-surgery
  The Health Questionnaire (EuroQoL EQ-5D) will be administered. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. The 5 areas that it measures include: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients | pre-operative
  Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath
Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients | 1 month post-surgery
  Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath
Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients | 3 months post-surgery
  Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath
Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients | 6 months post-surgery
  Edmonton Symptom Assessment Scale is a questionnaire used to rate the intensity of nine common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath
Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer | pre-operative
  Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer.
Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer | 1 month post-surgery
  Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer.
Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer | 3 months post-surgery
  Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer.
Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer | 6 months post-surgery
  Edmonton-33 is a patient reported outcomes measurement scale that was created by patients to measure the main functional areas of concern for patients with head and neck cancer.
Patient demographics including age, gender, T-stage, date of surgery | pre-operative
  Patient demographics including age, gender, T-stage, date of surgery: these variables will be entered into the Noona clinician portal by the research nurse
ER admissions related to aspiration pneumonia or dehydration | 6 month post surgery
  admissions related to aspiration pneumonia or dehydration: these will be entered into the Noona system by the research nurse, who will access Connect Care at the end of the 6-month period for each patient to record any such events

SECONDARY OUTCOMES:
Adherence to exercise using Mobili-T system | Up to 6 months, calculated from date of enrollment until the date of study completion or patient exit interview, whichever came first
  Adherence. Daily adherence logs are automatically collected by the Mobili-T system. Daily adherence as a percent of trials completed of those prescribed (e.g., 70/72*100) will be used to calculate average weekly adherence for each participant
Targets met when using Mobili-T system | Up to 6 months, calculated from date of enrollment until the date of study completion or patient exit interview, whichever came first
  Targets met: The daily percentage of exercise targets that the participant completes is automatically logged in the clinician portal.
Top three dysphagia symptoms reported on a weekly basis | Up to 6 months, calculated from date of enrollment until the date of study completion or patient exit interview, whichever came first
  Top three dysphagia symptoms reported on a weekly basis, where dysphagia symptoms include: coughing or choking, voice quality; food/liquid through nose; food/liquid out of mouth; watery eyes; food going down the wrong way; pain when swallowing; food felt stuck in throat; food felt stuck in cheeks; food in mouth after eating; long time to eat; reflux.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Rieger, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No